CLINICAL TRIAL: NCT03210675
Title: Early Detection and Treatment of Respiratory Sleep Disorders in Children With Down Syndrome
Acronym: RESPIRE21
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Hôpital Necker-Enfants Malades (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DP-TRS-T21
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Down Syndrome; Obstructive Sleep Apnea of Newborn
MeSH Terms: conditions — Down Syndrome | interventions — Polysomnography

STUDY DESIGN:
Intervention Model Description: Interventional, comparative, open label, multi-center study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Other): Will have a PSG at home every 6 months (± 1 month) from the age of 6 months until the age of 3 years.
  Interventions: Diagnostic Test: Polysomnography (PSG)
- Standard Care Group (Other): Will have a single PSG at home which will give a reference in the Down Syndrome population of 3 years old and will be used as reference to the study group
  Interventions: Diagnostic Test: Polysomnography (PSG)

INTERVENTIONS:
Diagnostic Test: Polysomnography (PSG) — PSG will be perfomed every 6 months in the Study group from the age of 6 months to 3 years

SUMMARY:
Interventional, comparative, open label, single-center study to demonstrate that an early (from 6 months of age) and systematic (every 6 months) screening of Obstructive Sleep Apnea (OSA) by polysomnography (PSG) in children with Down Syndrome during the first 3 years of life is associated with an improved neurocognitive development at the age of 3 years.

ELIGIBILITY:
Inclusion criteria :

Down Syndrome Age 6 months or less for the Study Group Age 30 to 36 months for the Standard Care Group Living in Paris or Paris area (75, 77, 78, 92, 93, 94, 95) Parents or legal representative agreeing with the study requirements and able to understand, date and sign the informed consent form before study enrollment French language is native mother tongue

Exclusion criteria :

Gestationnel age < 36 completed amenorrhoea weeks Patient who have or had acute CNS suffering signs Patients with Down Syndrome already had continuous positive airway pressure treatment for OSA Patients participating in another clinical study or for whom a participation to another biomedical research is expected before the end or their follow-up

Ages: 6 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean Griffith Mental Development Scale (GMDS) scores | At the age of 3 years
  Mean Griffith Mental Development Scale (GMDS) scores at the age of 3 years will be compared between the 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte FAUROUX, Professor, Study Chair — Hôpital Necker-Enfants Malade; Clotilde MIRCHER, Doctor, Principal Investigator — Institut Jérôme Lejeune
Locations (1):
- Institut Jérome Lejeune, Paris, France

REFERENCES:
- [Background] Lal C, White DR, Joseph JE, van Bakergem K, LaRosa A. Sleep-disordered breathing in Down syndrome. Chest. 2015 Feb;147(2):570-579. doi: 10.1378/chest.14-0266. PMID 25644910
- [Background] Bertrand P, Navarro H, Caussade S, Holmgren N, Sanchez I. Airway anomalies in children with Down syndrome: endoscopic findings. Pediatr Pulmonol. 2003 Aug;36(2):137-41. doi: 10.1002/ppul.10332. PMID 12833493
- [Background] Fricke BL, Donnelly LF, Shott SR, Kalra M, Poe SA, Chini BA, Amin RS. Comparison of lingual tonsil size as depicted on MR imaging between children with obstructive sleep apnea despite previous tonsillectomy and adenoidectomy and normal controls. Pediatr Radiol. 2006 Jun;36(6):518-23. doi: 10.1007/s00247-006-0149-7. Epub 2006 Apr 5. PMID 16596369
- [Background] Shires CB, Anold SL, Schoumacher RA, Dehoff GW, Donepudi SK, Stocks RM. Body mass index as an indicator of obstructive sleep apnea in pediatric Down syndrome. Int J Pediatr Otorhinolaryngol. 2010 Jul;74(7):768-72. doi: 10.1016/j.ijporl.2010.03.050. Epub 2010 May 7. PMID 20452066
- [Background] Marcus CL, Brooks LJ, Draper KA, Gozal D, Halbower AC, Jones J, Schechter MS, Ward SD, Sheldon SH, Shiffman RN, Lehmann C, Spruyt K; American Academy of Pediatrics. Diagnosis and management of childhood obstructive sleep apnea syndrome. Pediatrics. 2012 Sep;130(3):e714-55. doi: 10.1542/peds.2012-1672. Epub 2012 Aug 27. PMID 22926176
- [Background] Breslin J, Spano G, Bootzin R, Anand P, Nadel L, Edgin J. Obstructive sleep apnea syndrome and cognition in Down syndrome. Dev Med Child Neurol. 2014 Jul;56(7):657-64. doi: 10.1111/dmcn.12376. Epub 2014 Jan 29. PMID 24471822
- [Background] Bull MJ; Committee on Genetics. Health supervision for children with Down syndrome. Pediatrics. 2011 Aug;128(2):393-406. doi: 10.1542/peds.2011-1605. Epub 2011 Jul 25. PMID 21788214
- [Background] Ellis JM, Tan HK, Gilbert RE, Muller DP, Henley W, Moy R, Pumphrey R, Ani C, Davies S, Edwards V, Green H, Salt A, Logan S. Supplementation with antioxidants and folinic acid for children with Down's syndrome: randomised controlled trial. BMJ. 2008 Mar 15;336(7644):594-7. doi: 10.1136/bmj.39465.544028.AE. Epub 2008 Feb 21. PMID 18296460
- See also: Sponsor and site investigator — http://www.institutlejeune.org/
- See also: Site investigator for PSG evaluation — http://vnietsommeil.aphp.fr/